CLINICAL TRIAL: NCT02321319
Title: An Open-Label, Safety and Pharmacokinetic Study of Hydromorphone Hydrochloride Extended-Release Tablets (Once-Daily Hydromorphone) in Opioid-Tolerant Pediatric Subjects With Chronic Pain
Brief Title: Open-Label Safety and PK Study of ER Hydromorphone Tablets in Opioid-Tolerant Pediatric Chronic Pain Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision - product discontinued
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COV02520124
Record Dates: First submitted 2014-12-12; First posted 2014-12-22 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
Keywords: Pediatric
MeSH Terms: conditions — Chronic Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydromorphone HCl ER Tablets (Experimental): Participants receive Hydromorphone HCl ER Tablets (4-16 mg, based on standard conversion ratios for common opioids)
  Interventions: Drug: Hydromorphone HCl ER Tablets

INTERVENTIONS:
Drug: Hydromorphone HCl ER Tablets — Hydromorphone hydrochloride (HCl) extended release tablet
  Other Names: Exalgo, Jurnista

SUMMARY:
This pediatric study is designed to provide safety information, dosing guidelines, and a pharmacokinetic (PK) evaluation of once-daily hydromorphone hydrochloride (HCl) extended-release (ER) tablets in children with chronic painful conditions who are "opioid-tolerant" prior to enrollment under the Pediatric Research Equity Act (PREA) of 2003.

ELIGIBILITY:
Inclusion:

1. Male or female subjects aged 7 to 17 years.
2. Chronic cancer or noncancer pain (requiring around-the-clock opioid treatment) currently managed with stable dose of oral or injectable opioid corresponding to at least 6 mg of hydromorphone per day for at least 5 days prior to first dose.
3. Female subjects of child bearing potential must have negative serum pregnancy test result at Screening and Day 1. If sexually active must be surgically sterilized at least 12 months prior to Screening or use contraception at least 30 days prior to Screening and for the duration of study participation and for at least 30 days after the last dose of study drug.
4. Male subjects, with reproductive potential, who are sexually active must agree to use an acceptable method of contraception for the duration of the study.
5. Opioid-tolerant.
6. Subjects must have established a favorable response to opioid therapy in reducing pain.
7. Subjects must require a minimum dose of 4 mg (1 JURNISTA tablet) and a maximum dose of 16 mg (1 EXALGO tablet) after determining 66% of the converted dose of hydromorphone HCl per day from an established conversion table.
8. Able to swallow a whole tablet without breaking, crushing, chewing or dissolving.
9. Expected to require extended opioid treatment for at least 1 week.
10. Subjects must be able to communicate effectively with study personnel.
11. Subjects and parents/legal guardian must be able and willing to follow all protocol requirements and study restrictions.

Exclusion:

1. Life expectancy of less than 4 weeks.
2. History of allergy or any significant intolerance with opioid treatment or allergies to sulfites.
3. Currently using opioid (transcutaneous) analgesic patches.
4. History of drug or alcohol dependence.
5. History of renal, hepatic, cardiovascular, or respiratory conditions that would contraindicate participation in this study.
6. Plan to undergo a surgical procedure within 3 days of Day 1 and for the duration of subject participation in the study. Subjects undergoing minor surgical procedures (eg, central line insertion, biopsies) will be eligible for participation in the study.
7. Exhibit hemodynamic instability.
8. Have dysphagia, or difficulty swallowing whole tablets.
9. Narrowing of the digestive tract, Short gut syndrome, inflammatory bowel disease, peritonitis, cystic fibrosis, Meckel's diverticulum, or past GI surgery.
10. Hypothyroidism, Addison's disease, asthma (including exercise induced asthma) requiring daily inhalers, an enlarged prostate, epilepsy, low blood pressure, seizure disorder, high intracranial brain pressure, gallbladder problems, pancreatic disease, liver disease, or kidney disease.
11. Ileostomy or paralytic ileus.
12. Blood-product transfusion within 2 weeks of enrollment or expected to require transfusion during study.
13. Participated in a study with an investigational drug or device in the past 30 days prior to screening.
14. Known history of human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Mallinckrodt
Locations (3):
- United States (3):
  - Jackson Memorial Hospital, University of Miami, Miami, Florida
  - Medical Professional Clinical Research, Miami, Florida
  - Clinical Pharmacology Services, Inc., Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydromorphone HCl ER Tablets
Started | 5
Completed | 0
Not Completed | 5
Not completed — Product discontinued | 5

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone HCl ER Tablets
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: Hispanic | 5
  White: Non-hispanic | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Clinically significant changes in vital signs, pulse oximetry, and/or clinical laboratory assessments, were recorded as AEs
Time Frame: 28 days
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone HCl ER Tablets
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: 28 days, including a 3-week extension
Arm/Group | Hydromorphone HCl ER Tablets
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone HCl ER Tablets (N=5)
Itching (General disorders) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1)
Leukocytosis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT02321319/Prot_SAP_000.pdf